CLINICAL TRIAL: NCT02022358
Title: A Randomised, Cross-over Phase II Study to Investigate the Efficacy and Safety of Glucarpidase for Routine Use After High Dose Methotrexate in Patients With Bone Sarcoma
Brief Title: Will Glucarpidase After Methotrexate Treatment for Bone Sarcoma Lead to Fewer Side Effects and Reduce Chemotherapy Delays?
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment almost complete, has been slow and challenging
Sponsor: University College, London (Other)
Collaborators: Richard Scowcroft Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06/085
Record Dates: First submitted 2013-11-26; First posted 2013-12-27 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Osteosarcoma; Spindle Cell Sarcoma of Bone
Keywords: Osteosarcoma; Methotrexate; Glucarpidase; Mucositis
MeSH Terms: conditions — Osteosarcoma; Mucositis | interventions — glucarpidase; Methotrexate; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M (Active Comparator): Methotrexate (12 g/m2 x 1, intravenously) with standard folinic acid rescue
  In arm A patients will receive cycle M first followed by cycle GluM. Cycle M starts with course M1 on day 1 followed by course M2 planned for day 8. Cycle GluM starts with course GluM1 on day 1 followed by GluM2 planned for day 8. Cycle GluM will not start for a minimum of 14 days from the beginning of course M2, or until bone marrow, renal and hepatic functions have completely recovered and the patient is clinically ready to receive further chemotherapy .
  Interventions: Drug: Methotrexate; Drug: Folinic Acid
- GluM (Experimental): Methotrexate (12 g/m2 x 1, intravenously) with folinic acid and glucarpidase rescue (50 units/kg x 1, intravenously).
  In arm B, patients will receive cycle GluM first followed by cycle M. Cycle GluM starts with course GluM1 on day 1 followed by GluM2 planned for day 8.Cycle M starts with course M1 on day 1 followed by course M2 planned for day 8. Cycle M will not start for a minimum of 14 days from the beginning of course GluM2, or until bone marrow, renal and hepatic function have completely recovered and the patient is clinically ready to receive further chemotherapy
  Interventions: Drug: Glucarpidase; Drug: Methotrexate; Drug: Folinic Acid

INTERVENTIONS:
Drug: Glucarpidase — Glucarpidase rescue (50 units/kg x 1, intravenously)
  Other Names: Voraxaze
  Arms: GluM
Drug: Methotrexate — Methotrexate (12 g/m2 x 1, intravenously)
Drug: Folinic Acid — Folinic acid rescue 15mg/m2 four times daily adjusted according to methotrexate levels

SUMMARY:
Methotrexate is one of the most effective chemotherapy drugs in the treatment of osteosarcoma and some other types of bone sarcoma which are treated the same way as osteosarcoma. However, it frequently leads to sore mouth, tummy pain and increased risk of developing infections.

The investigators try to save or "rescue" normal cells from the side effects of methotrexate by giving a drug called folinic acid. Folinic acid is started 24 hours after methotrexate and given regularly until methotrexate levels are really low and not dangerous to normal cells anymore. Despite this rescue, side effects are still a problem and many patients are not well enough to receive subsequent chemotherapy on time. Almost half of the planned chemotherapy cycles are not given on time due to methotrexate side effects.

In this study the investigators will examine if adding a drug called glucarpidase to folinic acid is helpful. Glucarpidase is an enzyme that inactivates methotrexate in the blood stream. Lower methotrexate concentration in the blood stream leads to fewer side effects. The investigators would like to see if glucarpidase helps patients to have their chemotherapy on time, by reducing the side effects of methotrexate.

DETAILED DESCRIPTION:
In this study the patient will receive 4 courses of high-dose methotrexate. High-dose methotrexate is normally given at weekly intervals, in blocks of two.The first two courses will be given on weeks 1 & 2; the second two courses on weeks 4 & 5. Two courses will be given with folinic acid rescue (standard high-dose methotrexate), and the other two will be given with glucarpidase rescue as well as folinic acid. This will enable us to compare whether there is any difference in side effects with and without glucarpidase and also how quickly patients recover from them.

Half of the patients will receive standard high-dose methotrexate on weeks 1 & 2 and high-dose methotrexate with glucarpidase on weeks 4 & 5 (arm A) and half of the patients will first have high-dose methotrexate with glucarpidase on weeks 1 & 2 and then standard high-dose methotrexate on weeks 4 & 5 (arm B).

All patients receiving methotrexate have daily blood tests to monitor the levels of methotrexate in their body, and monitor their kidney function. However, patients on this study will have extra blood tests for chemotherapy drug levels and glucarpidase antibody levels. During each hospital admission for chemotherapy, blood samples will be taken as follows:

Day 1: Just before starting methotrexate (extra blood test) and at the end of methotrexate infusion (extra blood test) Day 2: 24 hours after starting methotrexate (routine blood test) and 20 minutes after the 24-hour blood test (i.e. just after the glucarpidase/placebo infusion) (extra blood test) Day 3+: Routine daily blood tests until the body has got rid of the methotrexate Extra blood samples will also be taken 15 days after starting each cycle and 1 month, 3 and 6 months, after starting the second cycle.

Patients will also be asked to complete mucositis assessment and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent from patient or parent/guardian Diagnosis of high grade osteosarcoma, localised or metastatic or high grade osteosarcoma as a second malignancy or spindle cell sarcoma of bone or relapsed high grade osteosarcoma Ability to comply with study and follow up procedures (WHO performance scale 0-2) No concomitant anti-cancer or investigational drugs during the study and complete resolution of toxicity related to previous treatment Life expectancy of at least 3 months Haematopoietic function: Absolute neutrophil count ≥1 x109/L, Platelets ≥75 x109/L Hepatic function: Bilirubin ≤1.5 x ULN Renal function: Glomerular Filtration Rate (radioisotope) ≥ 70 ml/min/1.73m2

Exclusion Criteria:

Previous treatment with glucarpidase Pregnant or breast feeding women (patients with reproductive potential of either gender must use contraception*) Concomitant treatment with agents which interact with methotrexate metabolism or excretion Serous effusions, including ascites and pleural effusions

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2007-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Estimate of the difference in proportions of patients ready to receive chemotherapy on Day 15 of each chemotherapy cycle comparing standard rescue and glucarpidase+standard rescue | Day 15 of each cycle
  The first day of each cycle is denoted Day 1. Therefore, the primary outcome will be the proportion of patients who are clinically fit to start cycle 2 of chemotherapy 14 days later.

SECONDARY OUTCOMES:
To investigate whether glucarpidase rescue after high-dose methotrexate reduces the incidence of methotrexate associated adverse effects | Day 8 and 15
  Incidence and grading of mucositis, renal toxicity, liver toxicity, neutropaenia, thrombocytopaenia and infections
Plasma methotrexate concentration | Every 24 hours from Time +24 until clearance of methotrexate
  Plasma methotrexate concentration
Incidence of glucarpidase related adverse effects | 6 weeks
  Each cycle lasts 3 weeks and patients receive two treatment cycles. The time frame will therefore be 6 weeks
Number of days required in hospital per cycle | 6 weeks
  Each cycle lasts 3 weeks and patients receive two treatment cycles. The time frame will therefore be 6 weeks
Assessment of quality of life | 6 weeks
  Completion of quality of life questionnaires at Day 1, 8, 15 each cycle
Serum anti-glucarpidase IgG levels following glucarpidase administration | 6 months
  Day 1, 8, 15 each cycle. Day 30 cycle 2, 3 and 6 months from entry
To investigate whether glucarpidase rescue after high-dose methotrexate reduces the severity of methotrexate associated adverse effects | Day 8 and 15
  Grading of mucositis, renal toxicity, liver toxicity, neutropaenia, thrombocytopaenia and infections
To investigate whether glucarpidase rescue after high-dose methotrexate reduces the duration of methotrexate associated adverse effects | Day 8 and 15
  Duration in days of mucositis, renal toxicity, liver toxicity, neutropaenia, thrombocytopaenia and infections
Plasma DAMPA concentration | Every 24 hours from Time +24 until clearance of methotrexate
  Plasma DAMPA concentration
Total dose of folinic acid rescue required per cycle | 6 weeks
  Each cycle lasts 3 weeks and patients receive two treatment cycles. The time frame will therefore be 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Whelan, Professor, Principal Investigator — University College London Hospitals
Locations (1):
- University College Hospital, London, United Kingdom